CLINICAL TRIAL: NCT05287672
Title: Retrospective Study of Effect of Adjuvant Chemoradiation of Gastric Carcinoma on Local Control and Survival
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Walaa Abdelshafy Ali, assistant lecrurer, Assiut University
Other Study IDs: 222
Record Dates: First submitted 2022-02-12; First posted 2022-03-18 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2022-03

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

SUMMARY:
Gastric cancer is the sixth most common cancer and the third most common cause of cancer-related death in the world.

The American Cancer Society estimates that about 26,560 cases of stomach cancer (16,160 in men and 10,400 in women) will be diagnosed in 2021. Median age at diagnosis is 68 years.

Decreases in gastric cancer have been attributed in part to widespread use of refrigeration. Other factors likely contributing to the decline in stomach cancer rates include lower rates of chronic Helicobacter pylori infection, thanks to improved sanitation and use of antibiotics, and increased screening in some countries.

Surgical resection is the principal therapy for gastric cancer, as it offers the only potential for cure.

Neoadjuvant chemotherapy has an established role in the management of gastric cancer. Perioperative chemotherapy, or postoperative chemotherapy plus chemoradiation, are preferred for localized gastric cancer. Because of lower toxicity, two-drug cytotoxic regimens are preferred for patients with advanced disease.

Adjuvant radiotherapy is associated with improvements in both overall and relapse-free survival and reductions in locoregional failure.

DETAILED DESCRIPTION:
Gastric cancer is the sixth most common cancer and the third most common cause of cancer-related death in the world.

The American Cancer Society estimates that about 26,560 cases of stomach cancer (16,160 in men and 10,400 in women) will be diagnosed in 2021. Median age at diagnosis is 68 years.

Decreases in gastric cancer have been attributed in part to widespread use of refrigeration. Other factors likely contributing to the decline in stomach cancer rates include lower rates of chronic Helicobacter pylori infection, thanks to improved sanitation and use of antibiotics, and increased screening in some countries.

Surgical resection is the principal therapy for gastric cancer, as it offers the only potential for cure.

Neoadjuvant chemotherapy has an established role in the management of gastric cancer. Perioperative chemotherapy, or postoperative chemotherapy plus chemoradiation, are preferred for localized gastric cancer. Because of lower toxicity, two-drug cytotoxic regimens are preferred for patients with advanced disease.

Adjuvant radiotherapy is associated with improvements in both overall and relapse-free survival and reductions in locoregional failure.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 to 70 years.
2. The World Health Organization Performance score 0-2.
3. Haemoglobin at least 10g/dl.
4. White blood cells at least 3000/mm3.
5. Platelets count at least 100000/mm3.
6. Bilirubin concentration no more than 25% higher than upper limit of normal .
7. Liver enzymes no greater than 2.5 times upper limit of normal.
8. Alkaline phosphatase no greater than 2 times upper limit of normal.
9. Creatinine concentration no more than 25% higher than the upper limit of normal .

Exclusion Criteria:

1. Second malignancy.
2. Prior abdominal irradiation.
3. Pregnant or nursing female.

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Gastric cancer is the sixth most common cancer and the third most common cause of cancer-related death in the world.
  Decreases in gastric cancer have been attributed in part to widespread use of refrigeration. Other factors likely contributing to the decline in stomach cancer rates include lower rates of chronic Helicobacter pylori infection, thanks to improved sanitation and use of antibiotics, and increased screening in some countries.
  Neoadjuvant chemotherapy has an established role in the management of gastric cancer. Perioperative chemotherapy, or postoperative chemotherapy plus chemoradiation, are preferred for localized gastric cancer. Because of lower toxicity, two-drug cytotoxic regimens are preferred for patients with advanced disease.
  Adjuvant radiotherapy is associated with improvements in both overall and relapse-free survival and reductions in locoregional failure.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2023-07 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Weight gain by BMI by kg/m2 | 2 years
  Weight gain by BMI by kg/m2